CLINICAL TRIAL: NCT04270799
Title: Lung Nodule Imaging Biobank for Radiomics and AI Research
Acronym: LIBRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: RM Partners West London Cancer Alliance (Unknown); Royal Brompton & Harefield NHS Foundation Trust (Other); University College London Hospitals (Other); Imperial College Healthcare NHS Trust (Other); Lewisham and Greenwich NHS Trust (Other Government); King's College Hospital NHS Trust (Other); Epsom and St Helier University Hospitals NHS Trust (Other); Institute of Cancer Research, United Kingdom (Other); Guy's and St Thomas' NHS Foundation Trust (Other); UCLH Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR5215
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer; Pulmonary Nodule, Multiple; Pulmonary Nodule, Solitary; Lung Neoplasms
Keywords: Incidental lung nodules; Radiomics; Artificial Intelligence; Machine Learning
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules; Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — CT scan images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Nodules: A cohort of 1000 patients with incidental lung nodules will be identified using clinical records at participating NHS sites.
  Link-anonymised CT scan images and data will be stored using a central database for radiomics and artificial intelligence research, to predict the risk of malignancy.
  Interventions: Diagnostic Test: Machine Learning Classification

INTERVENTIONS:
Diagnostic Test: Machine Learning Classification — Patient's scans will be used as input into in-house software to extract multiple radiomics features. These features will be used to develop a risk-signature which can predict malignancy risk. Patient scans will also be used as input into deep learning/convolutional neural network models to perform automated imaging classification.

SUMMARY:
This study will collect retrospective CT scan images and clinical data from participants with incidental lung nodules seen in hospitals across London. The investigators will research whether machine learning can be used to predict which participants will develop lung cancer, to improve early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Baseline CT thorax imaging reported as having pulmonary nodule(s) between 5 and 30mm in the last 10 years.
* Ground truth known (either scan data showing stability for 2 years (based on diameter) or one year (based on volumetry), complete resolution, or biopsy-proven malignancy.
* Slice thickness < 2.5mm.

Exclusion Criteria:

* • Absence of at least one technically adequate CT thorax imaging series (defined by visual inspection of presence of imaging data of the thorax in the DICOM record).

  * Slice thickness > 2.5mm.
  * Imaging > 10 years old.
  * Ground truth unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously identified lung nodules.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Development of an imaging biobank | 1 year
  The primary endpoint will be met if we are able to store baseline CT scans and the minimum clinical data set for 1000 patients.

SECONDARY OUTCOMES:
Discovery of a CT-thorax based radiomics profile to predict cancer risk. | 1 year
  We aim to identify distinct clusters of radiomics variables to generate a radiomics predictive vector (RPV), which can be used to stratify patients according to malignancy risk. This vector will be used in multivariate analysis and compared to existing risk models.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MBBS PhD, Study Chair — The Royal Marsden Hospital
Locations (5):
- United Kingdom (5):
  - Royal Marsden - Surrey, Sutton, England
  - Lewisham and Greenwich NHS Trust, London, Greater London
  - Epsom and St Helier's Hospitals NHS Trust, Carshalton, Surrey
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Brompton NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided